CLINICAL TRIAL: NCT05553171
Title: The Validity and Reliability of the Turkish Version of Brief Infant Sleep Questionnaire Revised (BISQ-R)
Brief Title: The Validity and Reliability of Brief Infant Sleep Questionnaire Revised (BISQ-R)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Perran Boran, Professor of Pediatrics, Marmara University
Other Study IDs: 02.09.2022.1127
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Insomnia; Behavioral Insomnia of Childhood
Keywords: insomnia; validity; Questionnaire
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brief Infant Sleep Questionnaire is a frequently used validated tool originally developed by Sadeh for evaluation of behavioral sleep problems in young children. It has been translated into Turkish and found reliable. The questionnaire has been revised and a norm referenced scoring system for the Brief Infant Sleep Questionnaire Revised (BISQ-R) was developed by Mindell and her team (Mindell JA, Gould RA, Tikotzy L, Leichman ES, Walters RM. Norm-referenced scoring system for the Brief Infant Sleep Questionnaire - Revised (BISQ-R). Sleep Med 2019; 63:106-114). We aimed to validate BISQ-R using exploratory and confirmatory factor analytical techniques, to provide evidence for its factor validity and reliability in a Turkish population.

DETAILED DESCRIPTION:
Brief Infant Sleep Questionnaire is a frequently used validated tool originally developed by Sadeh for evaluation of behavioral sleep problems in young children. It has been translated into Turkish and found reliable. The questionnaire has been revised and a norm referenced scoring system for the Brief Infant Sleep Questionnaire Revised (BISQ-R) was developed by Mindell and her team (Mindell JA, Gould RA, Tikotzy L, Leichman ES, Walters RM. Norm-referenced scoring system for the Brief Infant Sleep Questionnaire - Revised (BISQ-R). Sleep Med 2019; 63:106-114). We aimed to validate BISQ-R using exploratory and confirmatory factor analytical techniques, to provide evidence for its factor validity and reliability in a Turkish population.

The BISQ-R consists of 33 questions with 19 questions for scoring. There are 3 subscales including infant sleep, parent perception and parent behavior. The total and each subscale score ranges from 0 to 100. Total score is the average of the 3 subscale scores. Higher scores indicate better sleep quality, more positive perception of infant sleep, and parental behaviors that promote healthy and independent sleep.

Independent Turkish to English, and back translations were completed, and reviewed by BISQ-R team for consistency, and identified problems were resolved. The study is designed as a prospective observational study with an anticipated sample size of 300 children. An online google survey will be developed on the google platform securing data collection by a confidential log in system which can be filled out from smartphones, tablet or computer. For a test-retest reliability evaluation, a retest will be conducted in 100 participants with a 3 weeks interval between the administrations using Cronbach's alpha internal consistency coefficients, item analysis and test-retest method. The project has received Institutional Review Board (IRB) from Marmara University School of Medicine (02.09.2022.1127). After the data collection is completed, an application and an agreement form will be filled out and sent to BISQ-R team for scoring.

ELIGIBILITY:
Inclusion Criteria:

* Term born, typically developing children aged between 3 to 36 months and their parents

Exclusion Criteria:

* Having chronic diseases

Ages: 3 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Typically developing, term born, healthy children between 3 to 36 months of age and their parents
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Turkish Validation of the Brief Infant Sleep Questionnaire Revised (BISQ-R) Survey | Baseline
  Brief Infant Sleep Questionnaire-Revised (BISQ-R) Survey will be validated using exploratory and confirmatory factor analytical techniques
Turkish Reliability of the Brief Infant Sleep Questionnaire Revised (BISQ-R) Survey | Baseline
  Reliability will be examined by re-applying the questionnaire to 100 participants 3 weeks after the application of the questionnaire, using Cronbach's alpha internal consistency coefficients, item analysis and test-retest method.
Turkish Reliability of the Brief Infant Sleep Questionnaire Revised (BISQ-R) Survey | at 3 weeks
  Reliability will be examined by re-applying the questionnaire to 100 participants 3 weeks after the application of the questionnaire, using Cronbach's alpha internal consistency coefficients, item analysis and test-retest method.

SECONDARY OUTCOMES:
Protective factors index | baseline
  Brief Infant Sleep Questionnaire-Revised (BISQ-R) Survey total scores will be summed by the average of 3 subscale scores. Scores from each subscale and total score ranges from 0 to 100; higher scores indicate better sleep quality, more positive perception of infant sleep, and parental behaviors that promote healthy and independent sleep.
Subscale scores for each protective factors | baseline
  Brief Infant Sleep Questionnaire-Revised (BISQ-R) Survey subscale scores [infant sleep (IS) subscale, parental perception (PP), Parental Behavior (PB) subscales] will be computed. Higher scores indicate better sleep quality, more positive perception of infant sleep, and parental behaviors that promote healthy and independent sleep.In the infant sleep (IS) subscale, there are 5 questions about sleep patterns: sleep onset latency, number and duration of waking up at night, longest sleep duration, and total night sleep. In the parental perception (PP) subscale, there are 3 questions regarding the caregiver's perception of difficulty in bedtime, night sleep and general child sleep problems (Question 32,28,14). Eleven questions in the Parental Behavior (PB) subscale about sleep ecology, including routine consistency at bedtime, bedtime, parental behavior at sleep onset, and night awakenings.

IPD SHARING:
Plan to Share IPD: No
Requests for wider sharing of data (for example in response to publications about the study and willingness to share), will be addressed on a case-by-case basis. Any data sharing request will be made to investigators through a pre-defined data requisition form. This form will contain information about the applicant, institution, purpose of data request, study objectives, ethical clearance of the study, etc. Once a request has been made the data governance body will discuss if that request was appropriate; data will be released following signing of the data sharing agreement. The data will be stored on the Marmara University servers and not be deposited in any 'community' database.